CLINICAL TRIAL: NCT02717884
Title: Phase I/II Study of Sensitization of Non-M3 Acute Myeloid Leukemia (AML) Blasts to All-trans Retinoic Acid (ATRA) by Epigenetic Treatment With Tranylcypromine (TCP), an Inhibitor of the Histone Lysine Demethylase 1 (LSD1)
Brief Title: Study of Sensitization of Non-M3 AML Blasts to ATRA by Epigenetic Treatment With Tranylcypromine (TCP)
Acronym: TRANSATRA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Luebbert (Other)
Collaborators: University Hospital Freiburg (Other)
Responsible Party: Sponsor-Investigator, Michael Luebbert, Prof. Dr. med., University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00806 UKF
Record Dates: First submitted 2016-02-04; First posted 2016-03-24 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: AML; MDS; relapsed; trans-retinoic acid ATRA; epigenetic treatment; non-M3 AML blasts; tranylcypromine TCP; LSD1; refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Recurrence | interventions — Tranylcypromine; Tretinoin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TCP, ATRA, Cytarabine (Experimental): Phase I part:
  The rolling-six phase I design will be used to determine the MTD of TCP in combination with fixed-dose of ATRA and with fixed-dose AraC in patients with AML/MDS.
  Intervention: Four dose levels of TCP (20 mg, 40 mg**, 60 mg**, 80 mg** on days 1-28) will be examined in combination with ATRA (45 mg/m2 on days 10-28) and with fixed-dose AraC (40 mg on days 1-10) in the first cycle. In case of dose-limiting toxicity (DLT) on the starting level 1 of 20 mg a de-escalation to dose level of 10 mg (level -1) will be investigated.
  **TCP dose will be slowly increased to achieve the necessary dose level and slowly tapered off at the end of treatment
  Interventions: Drug: tranylcypromine; Drug: all-trans retinoic acid; Drug: cytarabine

INTERVENTIONS:
Drug: tranylcypromine — TCP p.o., daily either 20, 40**, 60**, 80** mg/day, (28d/cycle)
  **TCP doses will be slowly increased during cycle 1 and slowly decreased at end of treatment (for details see study protocol)
  Other Names: TCP; Jatrosom®
Drug: all-trans retinoic acid — 45mg/m2 (days 10-28), CAVE: ATRA will be administered without interruption until inclusively cycle 3. At the beginning of the cycle 4 a nine-day break corresponding to the first nine days of the AraC treatment will be performed, thereafter the ATRA-therapy will be continued with a nine-day interruption every fourth cycle. That means that the therapy in cycles 1, 4, 7, 10, 13 etc. In other cycles ATRA will be given without interruption
  Other Names: ATRA; Vesanoid®
Drug: cytarabine — 40mg s.c. (days 1-10)
  Other Names: Alexan®; AraC

SUMMARY:
The objective of the phase I part of the trial is the determination of the maximum tolerated dose (MTD) of TCP (Tranylcypromine) in combination with fixed-dose ATRA (all-trans-retinoic acid) and with fixed-dose AraC (Cytarabine) and to derive the recommended phase II dose (RP2D) in patients with non-APL AML or MDS for whom no standard treatment is available or who failed azanucleoside treatment.

The objective of the phase II part of the trial is a first evaluation of the efficacy of TCP at the RP2D in combination with fixed-dose ATRA and with fixed-dose AraC as basis for further investigations of TCP

DETAILED DESCRIPTION:
Study treatment: TCP + ATRA + AraC Four dose levels of TCP (20 mg, 40 mg, 60 mg, 80 mg on days 1-28) will be examined in combination with fixed dose ATRA (45 mg/m2 on days 10-28) and fixed-dose AraC (40 mg on days 1-10) in the first cycle.

In further cycles patients will be treated in the same manner, except for ATRA which will be administered continuously with a nine-day interruption at the beginning of every fourth cycle.

Follow-up per patient: Until twelve months after registration of the last patient.

Duration of intervention per patient: Until relapse/progression, unacceptable toxicity or until twelve months after registration of the last patient, whatever occurs first

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this trial must meet all of the following criteria:

1. Patients >18 years (no upper age limit);
2. AML (WHO) or intermediate or higher risk MDS/ Chronic Myelomonocytic Leukemia (CMML) (IPSS-R >3.0);
3. No standard treatment available (comorbidities, higher age, refractoriness to standard or salvage chemotherapy and allografting, azanucleosides failure*);
4. Patients with < 30.000 leukocytes/µl;
5. Eastern Cooperative Oncology Group (ECOG) 0,1,2;
6. Written informed consent obtained according to international guidelines and local laws;
7. Ability to understand the nature of the trial and the trial related procedures and to comply with them.

   * Azanucleosides failure is defined as 1) no response after at least three (AML) or six (MDS) cycles of azacitidine or decitabine, 2) disease progression under treatment or 3) grade 3-4 non-hematologic toxicity.

Exclusion Criteria:

Patients eligible for this trial must not meet any of the following criteria:

1. Acute promyelocytic leukemia (APL, French-American-British classification system (FAB) M3);
2. Eligibility for standard induction or consolidation chemotherapy, immediate allografting, or a hypomethylating agent;
3. AML with central nervous system (CNS) involvement;
4. AraC treatment within one month prior to registration;
5. Prior exposure to histone deacetylase inhibitors, including sodium valproate within one month prior to registration;
6. Stem cell transplant patient with graft-versus-host disease (GvHD) or under systemic immunosuppression;
7. Previous gastrointestinal surgery that might interfere with drug absorption;
8. Pheochromocytoma;
9. Carcinoid tumor;
10. Confirmed or suspected cerebrovascular disease;
11. Vascular malformations including aneurysm;
12. Severe renal insufficiency;
13. Severe or poorly controlled hypertension;
14. Severe cardiovascular disease;
15. Hepatic insufficiency/liver disease;
16. Porphyria;
17. Diabetes insipidus;
18. History or presence of malignant hyperthermia;
19. Known psychiatric disorders;
20. Known allergy against soy beans or peanuts;
21. Known hypersensitivity to or intolerance of one of the trial drugs or its constituents (e.g. lactose, corn starch, indigocarmine (TCP), corn starch (AraC), other retinoids (ATRA));
22. Simultaneous intake of the prohibited medication, incl. linezolid, that is likely to cause interactions (see detailed list study protocol);
23. Patients who refuse to follow study-specific dietary guidelines;
24. Known or persistent abuse of medication, drugs or alcohol;
25. Current or planned pregnancy, nursing period;
26. Failure to use safe methods of contraception;
27. Simultaneous participation in other interventional trials which could interfere with this trial and/or participation before the end of a required restriction period;
28. Participation in a clinical trial within the last 30 days before the start of this trial
29. Persons who are in a relationship of dependence/employment with the sponsor or the investigator;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
MTD determination of TCP in combination with fixed-dose of ATRA and with fixed-dose Cytarabine; | first 28 days of treatment
  MTD determination of TCP in combination with fixed-dose of ATRA and with fixed-dose Cytarabine;

SECONDARY OUTCOMES:
Objective best response | through study completion, an average of one year
  (CR complete remission, CRi complete remission with incomplete blood count recovery, PR partial remission)
Overall survival (OS) | 12 months
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lübbert, MD, Prof., Principal Investigator — Medical Center - University of Freiburg
Locations (6):
- Germany (6):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinik Düsseldorf, Medical School Duesseldorf, Düsseldorf
  - Universitätsklinikum Frankfurt Main, Medical School Frankfurt, Frankfurt am Main
  - Universitätsklinikum Freiburg, Medical School Freiburg, Freiburg im Breisgau
  - Klinikum München rechts der Isar, Medical School Munich rechts der Isar, München, Munich
  - Universitätsklinikum Tübingen, Medical School Tuebingen, Tübingen, Tuebingen

IPD SHARING:
Plan to Share IPD: No